CLINICAL TRIAL: NCT05651711
Title: A Phase 3, Randomized, 24-week, Placebo-controlled, Double-blind Study to Assess the Efficacy, Safety and Tolerability of Rocatinlimab (AMG 451) Monotherapy in Adult Subjects With Moderate-to-severe Atopic Dermatitis (AD) (ROCKET-Horizon)
Brief Title: A Study Assessing Rocatinlimab (AMG 451) Monotherapy in Moderate-to-severe Atopic Dermatitis (AD) (ROCKET-Horizon)
Acronym: ROCKET-Horizon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210143; 2022-501538-44 (Other: EU CT Number)
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; AMG 451; KHK 4083; Eczema; Rocatinlimab
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rocatinlimab (Experimental): Rocatinlimab Dose 1 every 4 weeks (Q4W) for 24 weeks with a loading dose at Week 2.
  Interventions: Drug: Rocatinlimab
- Placebo (Placebo Comparator): Placebo Q4W for 24 weeks with a loading dose at Week 2.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rocatinlimab — Rocatinlimab will be administered through a subcutaneous (SC) injection.
  Other Names: AMG 451; KHK 4083
  Arms: Rocatinlimab
Other: Placebo — The matching placebo will be administered through a SC injection.
  Arms: Placebo

SUMMARY:
The co-primary objectives of the study are to:

* Evaluate the efficacy of rocatinlimab compared with placebo at Week 24, assessed using Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD).
* Evaluate the efficacy of rocatinlimab compared with placebo at Week 24, assessed using Eczema Area and Severity Index (EASI).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (or ≥ legal adult age within the country if it is older than 18 years at signing of informed consent) with a diagnosis of AD according to the AAD Consensus Criteria (2014) present for at least 12 months
* History of inadequate response to TCS (Topical Corticosteroid) of medium or higher potency (with or without topical calcineurin inhibitors [TCI]) as appropriate or for whom topical treatments are otherwise medically inadvisable (eg, because of important side effects or safety risks).
* EASI score ≥16
* vIGA-AD score ≥3
* ≥10% body surface area (BSA) of AD involvement
* Worst pruritus numerical rating scale ≥ 4

Exclusion Criteria:

* Treatment with a biological product within 12 weeks or 5 half-lives, whichever is longer, prior to Day 1
* Treatment with any of the following medications or therapies within 4 weeks or 5 half-lives, whichever is longer, prior to Day 1:

  * Systemic corticosteroids
  * Systemic immunosuppressants
  * Phototherapy
  * Oral or topical Janus kinase inhibitors
* Treatment with any of the following medications or therapies within 1 week, prior to Day 1:

  * TCS of any potency
  * TCI
  * Topical phosphodiesterase type 4 (PDE4) inhibitors
  * Other topical immunosuppressive agents
  * Combination agents including TCS of any potency or TCI, PDE4 inhibitors, or other immunosuppressive agents

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Achievement of a Validated Investigator's Global Assessment for Atopic Dermatitis Score of 0 (Clear) or 1 (Almost Clear) with a ≥ 2 Point Reduction From Baseline (vIGA-AD 0/1) at Week 24 | Baseline and Week 24
Achievement of ≥ 75% Reduction From Baseline in EASI Score (EASI 75) at Week 24 | Baseline and Week 24

SECONDARY OUTCOMES:
Achievement of EASI 75 at Week 16 | Baseline and Week 16
Achievement of vIGA-AD 0/1 at Week 16 | Baseline and Week 16
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of Daily Worst Pruritus Numeric Rating Scale (NRS) Score at Week 16 in Participants with Baseline Weekly Average of Daily Worst Pruritus NRS Score ≥ 4 | Baseline and Week 16
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of Daily Worst Pruritus NRS Score at Week 24 in Participants with Baseline Weekly Average of Daily Worst Pruritus NRS Score ≥ 4 | Baseline and Week 24
Achievement of ≥ 90% Reduction From Baseline in EASI Score (EASI 90) at Week 24 | Baseline and Week 24
Achievement of ≥ 4-point Reduction From Baseline in Weekly Average of AD Skin Pain NRS Score at Week 24 in Participants with Baseline Weekly Average of AD Skin Pain NRS Score ≥ 4 | Baseline to Week 24
Achievement of vIGA-AD 1 Response With Presence of Only Barely Perceptible Erythema or vIGA-AD 0 Response (Revised Investigator's Global Assessment [rIGA] 0/1) at Week 24 | Baseline and Week 24
Achievement of a Facial AD Severity Score of Clear at Week 24 for Participants with Facial AD at Baseline | Baseline and Week 24
Achievement of a Hand AD Severity Score of Clear at Week 24 for Participants with Hand AD at Baseline | Baseline and Week 24
Change From Baseline in Weekly Average of Daily Worst Pruritus NRS Score at Week 16 | Baseline and Week 16
Change From Baseline in Weekly Average of Daily Worst Pruritus NRS Score at Week 24 | Baseline and Week 24
Change from Baseline in SCORing Atopic Dermatitis (SCORAD) Itch Visual Analogue Scale (VAS) Score at Week 16 | Baseline and Week 16
Change From Baseline in SCORAD Itch VAS Score at Week 24 | Baseline and Week 24
Achievement of a ≥ 4-point Reduction From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 24 in Participants with Baseline DLQI ≥ 4 | Baseline and Week 24
Change From Baseline in DLQI Score at Week 24 | Baseline and Week 24
Achievement of a ≥ 4-point Reduction From Baseline in Patient Oriented Eczema Measure (POEM) Score at Week 24 in Participants with Baseline POEM Score ≥ 4 | Baseline and Week 24
Change from Baseline in POEM Score at Week 24 | Baseline and Week 24
Achievement of ≥ 4-point Reduction from Baseline in Weekly Average of AD Skin Pain NRS Score at Week 16 in Participants with Baseline Weekly Average of AD Skin Pain NRS Score ≥ 4 | Baseline to Week 16
Change From Baseline in Weekly Average of Daily AD Skin Pain NRS Score at Week 24 | Baseline to Week 24
Change from Baseline in Weekly Average of Daily AD Skin Pain NRS Score at Week 16 | Baseline and Week 16
Achievement of ≥ 3-point Reduction from Baseline in Weekly Average of AD Skin Pain NRS Score at Week 24 in Participants with Baseline Weekly Average of AD Skin Pain NRS Score ≥ 3 | Baseline to Week 24
Achievement of ≥ 3-point Reduction from Baseline in Weekly Average of AD Skin Pain NRS Score at Week 16 in Participants with Baseline Weekly Average of AD Skin Pain NRS Score ≥ 3 | Baseline to Week 16
Change From Baseline in Weekly Average of Daily Sleep Disturbance NRS Score at Week 24 | Baseline to Week 24
Achievement of Hospital Anxiety and Depression Scale (HADS)-anxiety Subscale Score <8 at Week 24 in Participants with Baseline HADS-anxiety Subscale Score ≥ 8 | Baseline and Week 24
Achievement of HADS-depression Subscale Score <8 at Week 24 in Participants with Baseline HADS-depression Subscale Score ≥ 8 | Baseline and Week 24
Change From Baseline in HADS-anxiety Subscale Score at Week 24 | Baseline and Week 24
Change From Baseline in HADS-depression Subscale Score at Week 24 | Baseline and Week 24
Achievement of a ≥ 8.7-point Reduction From Baseline in SCORAD Score at Week 24 in Participants with Baseline SCORAD Score ≥ 8.7 | Baseline and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (197):
- United States (69):
  - Research Solutions of Arizona, PC, Litchfield Park, Arizona
  - Center for Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Clinical Trials Institute of Northwest Arkansas, Fayetteville, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Velocity Clinical Research Chula Vista, Chula Vista, California
  - West Coast Research LLC, Dublin, California
  - California Dermatology and Clinical Research Institute, Encinitas, California
  - Center for Dermatology Clinical Research Inc, Fremont, California
  - Velocity Clinical Research - San Diego, La Mesa, California
  - Velocity Clinical Research - North Hollywood, North Hollywood, California
  - Cura Clinical Research, Palmdale, California
  - University of California at San Francisco, Dermatology Clinic at Mount Zion, San Francisco, California
  - Clinical Science Institute, Santa Monica, California
  - Clarity Dermatology, Castle Rock, Colorado
  - Velocity Clinical Research - Denver, Denver, Colorado
  - Foxhall Research Center, Washington D.C., District of Columbia
  - Renaissance Research and Medical Group, Cape Coral, Florida
  - Driven Research LLC, Coral Gables, Florida
  - Saint Jude Clinical Research, Doral, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Glick Skin Institute, Margate, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Innovation Medical Research Center Inc, Palmetto Bay, Florida
  - University of South Florida Health Morsani Center for Advanced Healthcare, Tampa, Florida
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Sneeze, Wheeze, and Itch Associates, LLC, Normal, Illinois
  - The South Bend Clinic LLP, South Bend, Indiana
  - Options Research Group LLC, West Lafayette, Indiana
  - Dermatology and Skin Cancer Center of Overland Park, Overland Park, Kansas
  - DS Research, Louisville, Kentucky
  - Kentucky Advanced Medical Research LLC, Murray, Kentucky
  - MetroBoston Clinical Partners, Brighton, Massachusetts
  - Wendy Sadoff MD Dermatology PC, Farmington Hills, Michigan
  - Revival Research Institute LLC, Troy, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Advanced Dermatology of the Midlands, Omaha, Nebraska
  - James Del Rosso Dermatology Research, Las Vegas, Nevada
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Weiss Medical, Riverdale, New Jersey
  - Corning Center For Clinical Research, Horseheads, New York
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Crystal Run Healthcare, Monroe, New York
  - Ace Clinical Trials, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - OptiSkin Medical, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke South Durham, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Bernstein Clinical Research Center LLC, Cincinnati, Ohio
  - The Ohio State University Dermatology East, Gahanna, Ohio
  - Velocity Clinical Research - Grants Pass, Grants Pass, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Asthma and Allergy Physicians of Rhode Island Clinical Research Institute, Warwick, Rhode Island
  - Bellaire Dermatology Associates, Bellaire, Texas
  - US Dermatology Partners Cedar Park, Cedar Park, Texas
  - Alina Clinical Trials, LLC, Dallas, Texas
  - Zenos Clinical Research, LLC, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - MedCare Pharma - Houston, Houston, Texas
  - FMCScience LLC, Lampasas, Texas
  - Epic Clinical Research Incorporated, Lewisville, Texas
  - Sienna Dermatology Research, Missouri City, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Andante Research, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - University of Utah MidValley Dermatology, Murray, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - MultiCare Institute for Research and Innovation, Spokane, Washington
- Australia (7):
  - St George Dermatology and Skin Cancer Centre, Darlinghurst, New South Wales
  - Premier Specialists, Kogarah, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Skin Health Institute, Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Belgium (3):
  - Hopital Erasme, Brussels
  - Clinique Andre Renard, Herstal
  - Dermatologie Maldegem, Maldegem
- Brazil (3):
  - CETI - Centro de Estudo em Terapias Inovadoras, Curitiba, Paraná
  - Centro Multidisciplinar de Estudos Clinicos - CEMEC, São Bernardo do Campo, São Paulo
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, São Paulo
- Canada (11):
  - Beacon Dermatology, Calgary, Alberta
  - Doctor Chih-Ho Hong Medical Incorporated, Surrey, British Columbia
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - The Centre for Clinical Trials Inc, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - XLR8 Medical Research, Incorporated, Windsor, Ontario
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Quebec
  - Clinique Dermatologique de Sherbrooke, Sherbrooke, Quebec
- Czechia (9):
  - Kozni ambulance Kutna Hora sro, Kutná Hora
  - Nemocnice Novy Jicin as, Nový Jičín
  - CCR Czech as, Pardubice
  - Fakultni nemocnice Plzen, Pilsen
  - Kozni ambulance Fialova sro, Prague
  - Dermamedest sro, Prague
  - CCR Prague sro, Prague
  - Praglandia sro, Prague
  - Dermatologicka ambulance MUDr Petr Trestik, Svitavy
- Denmark (2):
  - Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Clinical Research Centre, Tartu
- Finland (4):
  - CRST Helsinki, Helsinki
  - CRST Turku, Helsinki
  - Oulun Yliopistollinen sairaala (OYS), Oulu
  - Terveystalo Tampere, Tampere
- Germany (11):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Hautzentrum Friedrichshain - Dermatologie, Berlin
  - Clinical Research Services Berlin GmbH, Berlin
  - Klinikum der Medizinischen Fakultaet der Martin-Luther-Universitaet Halle-Wittenberg, Halle
  - Dermatologikum Hamburg, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Velocity Clinical Research, Leipzig
  - Universitaetsklinikum Muenster, Münster
  - KliFOs Klinische Forschung Osnabrueck, Osnabrück
  - Hautarztpraxis Mortazawi, Remscheid
  - Helios Klinikum Wuppertal, Wuppertal
- Japan (15):
  - Miyata Dermatology Clinic, Matsudo-shi, Chiba
  - International University of Health and Welfare Narita Hospital, Narita-shi, Chiba
  - Kobe University Hospital, Kobe, Hyōgo
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - National Hospital Organization Sagamihara National Hospital, Sagamihara-shi, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Osaka Habikino Medical Center, Habikino-shi, Osaka
  - Dermatology and Ophthalmology Kume Clinic, Sakai-shi, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Mita Dermatology Clinic, Minato-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Seibo International Catholic Hospital, Shinjuku-ku, Tokyo
  - Sugamo Kobayashi Derma Clinic, Toshima-ku, Tokyo
  - Shirasaki Dermatology Clinic, Takaoka-shi, Toyama
- Mexico (3):
  - Clínica de Enfermedades Crónicas y de Procedimientos Especiales, Morelia, Michoacán
  - Scientia Investigacion Clinica Sc, Chihuahua City
  - Phylasis Clínicas Research S. De R. L. De C. V., Cuautitlán Izcalli
- Poland (10):
  - ClinicMed Daniluk Nowak Spolka komandytowa, Bialystok
  - Dermapolis Medical Dermatology Center dr n med Edyta Gebska, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centermed krakow sp zoo, Krakow
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - AppleTreeClinics Network Spzoo, Lodz
  - Amicare Spolka z ograniczona odpowiedzialnoscia Spolka Komandytowa Amicare Centrum Medyczne, Lodz
  - Clinical Best Solutions Sp zoo Spolka Komandytowa, Lublin
  - Clinical Research Center Spzoo Medic-R Spolka Komandytowa, Poznan
  - Evimed sp zoo centrum medyczne evimed, Warsaw
- Portugal (5):
  - Hospital Garcia de Orta, EPE, Almada
  - Centro Hospitalar e Universitario de Coimbra, EPE, Coimbra
  - Hospital Cuf Descobertas, Lisbon
  - Centro Hospitalar Universitario do Porto, EPE - Hospital de Santo Antonio, Porto
  - Centro Hospitalar de Sao Joao EPE - Hospital de Sao Joao, Porto
- Spitalul Clinic Colentina, Bucharest, Romania
- South Africa (3):
  - Ryexo Clinical Research, Centurion, Gauteng
  - About Allergy, Johannesburg, Gauteng
  - Hiway Medical Centre, Durban
- South Korea (20):
  - Korea University Ansan Hospital, Ansansi, Gyeonggido
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chosun University Hospital, Gwangju
  - The Catholic University of Korea Incheon St Marys Hospital, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - National Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Asan Medical Center, Seoul
  - The Catholic Univ of Korea Seoul St Marys Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Ajou University Hospital, Suwon-si, Gyeonggi-do
- Spain (8):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital de Manises, Manises, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia, Valencia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
- Karolinska Universitetssjukhuset Solna, Stockholm, Sweden
- Turkey (Türkiye) (7):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Gaziantep Universitesi Tip Fakultesi Hastanesi, Gaziantep
  - Bezmialem Vakif Universitesi Hastanesi, Istanbul
  - Bakircay Universitesi Cigli Egitim ve Arastirma Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Sakarya Egitim ve Arastirma Hastanesi, Sakarya
- United Kingdom (3):
  - Lakeside Healthcare, Corby
  - Guys Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Guttman-Yassky E, Kabashima K, Worm M, Luna PC, Hong HC, Chovatiya R, Bernstein JA, Kern JS, Ehst BD, Magnolo N, Herranz-Pinto P, Stein Gold L, Sofen H, Pink AE, Esfandiari E, Arai T, Yang Y, Shi R, Barragan C, Kricorian G, Schwartz-Sagi L, Bissonnette R. Efficacy and safety of rocatinlimab for the treatment of moderate-to-severe atopic dermatitis in ROCKET-IGNITE and ROCKET-HORIZON: two global, double-blind, placebo-controlled, randomised phase 3 clinical trials. Lancet. 2026 Jan 3;407(10523):53-66. doi: 10.1016/S0140-6736(25)01865-3. Epub 2025 Nov 25. PMID 41314226
- [Derived] Guttman-Yassky E, Simpson E, Bissonnette R, Eichenfield LF, Kabashima K, Luna PC, Hercogova JT, Spelman L, Worm M, Esfandiari E, Arai T, Mano H, Charuworn P, Wang A, Kricorian G. ROCKET: a phase 3 program evaluating the efficacy and safety of rocatinlimab in moderate-to-severe atopic dermatitis. Immunotherapy. 2025 Feb;17(2):83-94. doi: 10.1080/1750743X.2025.2464528. Epub 2025 Feb 26. PMID 40012373
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com